CLINICAL TRIAL: NCT04123756
Title: Smerteprofiler Som Redskab Til at prædiktere Effekten af 6-8 Ugers GLA:D®-forløb Hos Patienter Med Smertefuld Slidgigt i knæene
Brief Title: Predicting Outcome Following Standardized Exercise Therapy in Knee Osteoarthritis Patients
Status: Terminated | Type: Observational
Why Stopped: Recruitment issues due to the corona virus and lack of funding to continue
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Kristian Kjær Petersen, Associate Professor, M.Sc., Ph.D., Aalborg University
Other Study IDs: N-20190045
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: standardized exercise therapy for knee OA patients — Standardized exercise therapy for 6-8 weeks (two times per week).

SUMMARY:
Pain sensitization has been associated with pain severity in people with knee osteoarthritis (KOA) and a neuropathic pain component has been identified in up to 30% of KOA patients. Mechanistic pain profiling aims to identify the underlying mechanisms in the peripheral and central nervous systems, which are associated to the clinical pain.

In addition, the mechanisms underlying the pain relieving effect of standardized exercise therapy are largely unknown, but it is hypothesized that they are linked to the patient's ability to activate the descending pain inhibitory pathways (conditioned pain modulation, CPM) in the central nervous system. Mechanistic pain profiling including CPM have been used prognostic to identify responders to treatment, but these measures as a prognostic tool for standardized exercise therapy has not been investigated.

The primary aim of this study is to investigate if mechanistic pain profiling alone or in combination with clinical pain measures before standardized exercise therapy can predict the patients' pain reduction following the exercise therapy program

ELIGIBILITY:
Inclusion Criteria:

* The American College of Rheumatology for clinical knee osteoarthritis (excluding radiological OA assessment)

Exclusion Criteria:

* Known factors to influence pain and pain sensitization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 patients with knee osteoarthritis scheduled for standardized exercise therapy
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
pain reduction | 1-2 weeks after last exercise session
  Pain measured on a numerical rating scale from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- FysioDanmark Aarhus, Aarhus, Denmark